CLINICAL TRIAL: NCT02269306
Title: Visceral Fat Area and Other Predictors of Ovarian Response During Clomiphene Citrate Ovulation Induction in Patients With Polycystic Ovary Syndrome
Brief Title: Predictors of Ovarian Response During Clomiphene Citrate Ovulation Induction in Patients With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia Obstetrics and Gynecology Group (Other)
Responsible Party: Principal Investigator, Dr Hamed Ellakwa, Dr Hamed Ellakwa, Menoufia Obstetrics and Gynecology Group
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Menoufia OGG-1
Record Dates: First submitted 2014-10-02; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Anovulation
Keywords: PCOS; clomiphene citrate; AMH; visceral fat area; HOMA-IR
MeSH Terms: conditions — Anovulation | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- clomiphen citrate(cc) (Experimental): Initial CC doses were 50 mg daily for 5 days starting on cycle day 3. In the case of an absent response, doses were increased to 100 and 150 mg daily in subsequent cycles.
  Interventions: Drug: clomiphen citrate

INTERVENTIONS:
Drug: clomiphen citrate — The study was carried out on 150 patients with PCOS. Initial clomiphen citrate (CC) doses were 50 mg daily for 5 days starting on cycle day 3. In the case of an absent response, doses were increased to 100 and 150 mg daily in subsequent cycles. First ovulation with CC was used as the end point.
  Other Names: clomid

SUMMARY:
The purpose of this study is to determine whether Visceral fat area and other criteria assessed during initial screening could predict the response to ovulation induction with clomiphene citrate (CC) in patients with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
The study was carried out on 150 patients with PCOS. Initial CC doses were 50 mg daily for 5 days starting on cycle day 3. In the case of an absent response, doses were increased to 100 and 150 mg daily in subsequent cycles. First ovulation with CC was used as the end point.Statistical methods Distribution of characteristics in patients is presented as the mean ± SD. We used the Mann-Whitney U test for exploratory comparison of initial parameters between responders and nonresponders. The univariate and multivariate relation with response to CC was assessed using logistic regression analysis. Backward stepwise elimination was used for the multivariate logistic analysis of prediction of patients being CRA, and P < 0.10 was used as a cut-off level for elimination of non-significant predictors from the prognostic model. The area under the receiver operating characteristics (ROC) curve (AUC) was used to assess the discriminative ability of the logistic models. SPSS with statistical package version 17 (SPSS Inc., Chicago, IL) and MedCalc Software version 12.4, (Ostend, Belgium) were employed for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* The study included 150 infertile women(age from 18 to 40 years) with PCOS diagnosed by the presence of at least two of the following [15]:

  1. Clinical hyperandrogenism: Hirsutism or acne vulgaris and/or biochemical hyperandrogenism (total testosterone >88 ng/dl or DHEAS >275 ug/dL)[16]. (2) Menstrual and/or ovulatory disturbances, mainly oligomenorrhea (interval between vaginal bleeding >35 days and < 6 months) or amenorrhea (bleeding interval >6 months). (3) Polycystic ovaries as visualized by transvaginal ultrasound (either 12 or more follicles measuring 2-9 mm in diameter or increased ovarian volume >10 cm3).

Exclusion Criteria:

* Patients having one or more of these criteria were excluded; Age <18 years or >40 years, body mass index (BMI) <18.5 kg/m2 or >35 kg/m2, pregnancy, endocrine disorders, systemic disease, current or previous (within the last 3 months) use of oral contraceptives, glucocorticoids, antiandrogens, ovulation induction or dopaminergic agents, use of antidiabetes, antiobesity drugs or history of tubal or ovarian surgery.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
ovulation | 3 months ( cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Hamed El Ellakwa, MD, Principal Investigator — Menoufiya faculty of medicine,menoufiya university,ministry of higher education
Locations (1):
- Menoufia University hospital, Shebin Elkom, Menoufia, Egypt

REFERENCES:
- [Derived] Ellakwa HE, Sanad ZF, Hamza HA, Emara MA, Elsayed MA. Predictors of patient responses to ovulation induction with clomiphene citrate in patients with polycystic ovary syndrome experiencing infertility. Int J Gynaecol Obstet. 2016 Apr;133(1):59-63. doi: 10.1016/j.ijgo.2015.09.008. Epub 2015 Dec 17. PMID 26848057